CLINICAL TRIAL: NCT03026010
Title: Early Detection of Central Blood Pressure and Arterial Stiffness (Pulse Wave Analysis) Can be a Predictor of Gestational Hypertension/Preeclampsia.
Brief Title: Central Blood Pressure
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Laura Vricella, MD, Principal investigator, St. Louis University
Other Study IDs: 23621
Record Dates: First submitted 2017-01-12; First posted 2017-01-20 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: central blood pressure — SphygmoCor XCEL will be used to measure both standard blood pressure in the arm and central pressure, the blood pressure at the heart.

SUMMARY:
The aim of the study is to check standard screening blood pressure in the arm and central blood pressure, the blood pressure at the heart in pregnant women. The standard brachial pressure is routinely monitored throughout pregnancy, however it is not sensitive enough to distinguish preeclampsia from other types of hypertension or to predict preeclampsia in those at risk. Central aortic pressure monitoring has become a valuable clinical tool and preliminary studies suggest that measuring of central blood pressure may be better predictor of preeclampsia. It is non invasive and doesn't require undressing. It involves using a standard blood pressure cuff placed around the thigh, checking carotid pulse and pressure with an ultrasound and taking measurements of the person neck to torso. With this knowledge it will be a useful screening tool to identify these patients at higher risk and hopefully lead to closer monitoring, earlier treatment and reduced morbidity and mortality

DETAILED DESCRIPTION:
When blood pressure is measured conventionally over the brachial artery it is assumed that these measurements accurately reflect pressures in the central circulation. However, central aortic pressure is the blood pressure at the root of aorta and are determined not only by cardiac output and peripheral vascular resistance, but by the stiffness of conduit arteries and the timing and magnitude of pressure wave reflection.

Studies have shown the importance of central aortic pressure and its implications in assessing the efficacy of antihypertensive treatment with respect to cardiovascular risk factors. In the CAFE Study the traditional method of measuring blood pressure in the arms has been shown to underestimate the efficacy of drugs such as amlodipine and overestimate the efficacy of those like atenolol (4). This clinical trial demonstrated that different medications for lowering blood pressure have different effects on the central aortic pressure and blood flow characteristics, despite producing similar brachial blood pressure readings. They also were able to show that central aortic pressures are a better independent predictor of cardiovascular and renal outcome. The Strong Heart Study went further to depict how central pressure are more predictive of the load imposed on the coronary and cerebral arteries and thereby bear a stronger relationship to vascular damage and prognosis.

Hypertensive disorders of pregnancy, in particular, preeclampsia, are a leading cause of maternal and neonatal morbidity and mortality. In the United States and the United Kingdom, approximately 5% of pregnancies are complicated by preeclampsia, and of these patients, 1-2% progress to eclampsia. It is estimated that these rates are higher in developing countries. An estimated 50,000 women die annually from preeclampsia worldwide. The presence of hypertension during pregnancy is also associated with a two-fold increase in the risk of gestational diabetes mellitus. In addition, a history of preeclampsia increases a women's subsequent risk of vascular disease, including hypertension, ischemic heart disease, myocardial infarction and stroke. The increased risk of complications is not limited to the mother; babies of women with hypertensive disorders during pregnancy are more likely to suffer adverse outcomes than those of women without hypertension. A large cross-sectional study observing more than 250,000 women and their infants showed that women with gestational hypertension were at a 30% greater risk of death or major morbidity, and women with pre-eclampsia had a 400% increased risk, compared to women without hypertension. Although preeclampsia is not preventable, early diagnosis, careful monitoring and aggressive treatment is crucial in preventing mortality.

The brachial pressure is routinely monitored throughout pregnancy, however it is not sensitive enough to distinguish preeclampsia from other types of hypertension or to predict preeclampsia in those at risk. Central aortic pressure monitoring has become a valuable clinical tool outside of pregnancy, particular in assessment of patient's hypertension, renal disease and diabetes. Preliminary studies suggest that measuring of central blood pressure may be predictive preeclampsia. In normal pregnancy aortic stiffness has been shown to vary throughout the pregnancy, reaching its lowest point in second trimester and rising again in the third trimester. A number of studies have investigated the change in pulse wave indices in the third trimester across the spectrum of hypertensive disorders. Central pressures, along with Augmentation pressure were found to be significantly higher in gestational hypertension and preeclampsia compared to normal pregnancy. In addition, Aortic augmentation pressure and pulse wave velocity has been shown to vary between preeclampsia, gestational hypertension, and normal pregnancy. The ability to accurately identify women at risk for preeclampsia would have significant clinical benefits. The ability to distinguish between hypertensive disorders and identify those women who have increased risk of preeclampsia can lead to better management of hypertensive disorders during pregnancy and therefore better outcomes for both mother and child. The aim of our study is to examine if early evaluation of central blood pressure and arterial stiffness (pulse wave analysis) can be a predictor of gestational hypertension/preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* ≤20 weeks pregnant

Exclusion Criteria:

* Multi-pregnancy; Fetal anomalies

Ages: 14 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant women > or equal to 14 year old to 60 years old
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
pulse wave analysis | 1 year
  pulse wave analysis can be a predictor of gestational hypertension/preeclampsia.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Vricella, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No